CLINICAL TRIAL: NCT00559637
Title: Single-arm, Open Study to Investigate the Efficacy, Safety and Tolerability of Monthly Subcutaneously Administered C.E.R.A. in Patients With Renal Anemia Not Yet Subject to Dialysis and Not Yet Permanently Treated With ESAs
Brief Title: A Study of Subcutaneous Mircera in Participants With Chronic Kidney Disease Not Treated With ESA or on Dialysis
Acronym: MERCUR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20888; 2007-000126-46 (EudraCT Number)
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (1):
- Methoxy polyethylene glycol-epoetin beta (Experimental): Methoxy polyethylene glycol-epoetin beta will be administered subcutaneously once a month. The starting dose will be 1.2 mcg/kg of body weight. Further dose adjustments will be performed during the study depending on the hemoglobin value. Total duration of treatment will be 9 months for all participants in the study and up to 11 months for participants who will be shifted to the dialysis.
  Interventions: Drug: Methoxy polyethylene glycol-epoetin beta

INTERVENTIONS:
Drug: Methoxy polyethylene glycol-epoetin beta — Methoxy polyethylene glycol-epoetin beta will be administered subcutaneously once a month. The starting dose will be 1.2 mcg/kg of body weight. Further dose adjustments will be performed during the study depending on the hemoglobin value. Total duration of treatment will be 9 months for all participants in the study and up to 11 months for participants who will be shifted to the dialysis.
  Other Names: Mircera

SUMMARY:
This single arm study will assess the efficacy and safety of subcutaneous Mircera for correction of anemia in participants with chronic kidney disease who are not treated with erythropoiesis stimulating agent (ESA) and not on dialysis. Eligible participants will receive Mircera by monthly subcutaneous injections. The initial dose, based on body weight, will be 1.2 micrograms/kilogram (mcg/kg). The anticipated time on study treatment is 9-11 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* chronic renal anemia;
* hemoglobin value less than or equal to (<=) 10.5 grams/deciliter (g/dL).

Exclusion Criteria:

* prior ESA therapy during previous 3 months;
* acute or chronic bleeding requiring therapy during previous 2 months;
* transfusion of red blood cells during previous 2 months;
* active malignant disease (except non-melanoma skin cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (47):
- Germany (47):
  - Ansbach
  - Arnsberg
  - Bad Aibling
  - Berlin
  - Bischofswerda
  - Bonn
  - Cologne
  - Dieburg
  - Dortmund
  - Düsseldorf
  - Emsdetten
  - Frankfurt
  - Friedberg
  - Grimma
  - Hamburg
  - Heidelberg
  - Hilden
  - Homburg
  - Hoyerswerda
  - Jena
  - Kaiserslautern
  - Loerrach
  - Ludwigslust
  - Lübeck
  - Lünen
  - Mainz
  - Malente
  - Mettmann
  - Mühlacker
  - München
  - Regensburg
  - Rheine
  - Saarlouis
  - Schwandorf in Bayern
  - Schweinfurt
  - Sindelfingen
  - Sinsheim
  - Tangermünde
  - Trier
  - Tübingen
  - Ulm
  - Velbert
  - Wetzlar
  - Wiesloch
  - Worms
  - Würzburg
  - Zwickau

RESULTS

PARTICIPANT FLOW:
Groups:
- Methoxy Polyethylene Glycol-epoetin Beta: Methoxy polyethylene glycol-epoetin beta was administered subcutaneously once a month. The starting dose was 1.2 micrograms per kilogram (mcg/kg) of body weight. Further dose adjustments were performed during the study depending on the hemoglobin value. Total duration of treatment was 9 months for all participants in the study and up to 11 months if participants were shifted to dialysis.
Period: Overall Study
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Started | 184
Completed | 130
Not Completed | 54
Not completed — Adverse Event | 22
Not completed — Withdrawal by Subject | 4
Not completed — Protocol Violation | 6
Not completed — Withdrawal criteria fulfilled | 4
Not completed — Failure to return | 6
Not completed — Insufficient response | 3
Not completed — Started requiring dialysis after month 7 | 2
Not completed — Suspected lung cancer | 1
Not completed — Participation in another study | 1
Not completed — Delayed administration of C.E.R.A | 1
Not completed — Change of center | 1
Not completed — Change of home | 1
Not completed — Inclusion or exclusion criteria violated | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of study medication.
Groups:
- Methoxy Polyethylene Glycol-epoetin Beta: Methoxy polyethylene glycol-epoetin beta was administered subcutaneously once a month. The starting dose was 1.2 mcg/kg of body weight. Further dose adjustments were performed during the study depending on the hemoglobin value. Total duration of treatment was 9 months for all participants in the study and up to 11 months if participants were shifted to dialysis.
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (15.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 93

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Both Hemoglobin Values of the Evaluation Phase in the Range of 11-12 Grams Per Deciliter (g/dL)
Description: Participants with both hemoglobin values of the evaluation phase (Months 8 and 9, i.e., Study Days 200-260, values were at least 21 days apart) in the range of 11-12 g/dL were classified as responder. Participants who received transfusion of erythrocytes between Study Day 139 and 260, or with at least one value missing or outside the range were classified as non-responder for the hemoglobin-range concerned.
Time Frame: Evaluation phase (Months 8 and 9)
Population: Intent to treat (ITT) population included all participants who received at least one dose of study medication with at least one hemoglobin value measured during treatment period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 178
percentage of participants | 10.67 [6.55 to 16.17]

2. Primary Outcome: Percentage of Participants With Both Hemoglobin Values of the Evaluation Phase in the Range of 11-13 g/dL
Description: Participants with both hemoglobin values of the evaluation phase (Months 8 and 9, i.e., Study Days 200-260, values were at least 21 days apart) in the range of 11-13 g/dL were classified as responder. Participants who received transfusion of erythrocytes between Study Day 139 and 260, or with at least one value missing or outside the range were classified as non-responder for the hemoglobin-range concerned.
Time Frame: Evaluation phase (Months 8 and 9)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 178
percentage of participants | 29.21 [22.65 to 36.48]

3. Secondary Outcome: Duration of Hemoglobin Values in the Range of 11-12 g/dL
Description: The duration of hemoglobin values staying within the range of 11-12 g/dL was defined as the number of (not necessarily consecutive) months with all corresponding hemoglobin values in the respective range. All months with missing hemoglobin values were counted as months where the hemoglobin value did not stay within the respective range.
Time Frame: Baseline to Month 9
Population: ITT population
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 178
months | 2.40 (1.796)

4. Primary Outcome: Change From Baseline in Hemoglobin Value to the Evaluation Phase
Description: The change from the baseline hemoglobin value to the mean hemoglobin value of the evaluation phase was only calculated if both the baseline value and the mean of the evaluation phase (mean of Months 8 and 9) were available. In case of only one available hemoglobin value within the evaluation phase, that single value replaced the mean.
Time Frame: Baseline, evaluation phase (Months 8 and 9)
Population: ITT population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 131
g/dL | 1.6 (1.10)

5. Secondary Outcome: Duration of Hemoglobin Values in the Range of 11-13 g/dL
Description: The duration of hemoglobin values staying within the range of 11-13 g/dL was defined as the number of (not necessarily consecutive) months with all corresponding hemoglobin values in the respective range. All months with missing hemoglobin values were counted as months where the hemoglobin value did not stay within the respective range.
Time Frame: Baseline to Month 9
Population: ITT population
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 178
months | 3.62 (2.450)

6. Secondary Outcome: Time to Increase of Hemoglobin Value to Over 11 g/dL
Description: The duration (number of months) until the hemoglobin value exceeded 11 g/dL for the first time was summarized for participants for whom at least one measured hemoglobin value exceeded 11 g/dL.
Time Frame: Baseline to Month 9
Population: ITT population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 152
months | 2.28 (1.649)

7. Secondary Outcome: Total Number of Dose Adjustments
Description: A dose adjustment was defined as a change versus the preceding dose. It included dose increase, dose reduction and dose interruption. An interruption (no dose given) was always counted as a dose adjustment, regardless of whether or not at the previous time point a dose had been administered. After an interruption a change in the dose relative to the dose given before the interruption was counted as a dose adjustment.
Time Frame: Baseline until Month 8
Population: ITT population
Measure: Number; unit: dose adjustments
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 178
dose adjustments
  Total number of dose adjustments | 595
  Total number of dose increases | 249
  Total number of dose reductions | 210
  Total number of dose interruptions | 136

8. Secondary Outcome: Total Number of Red Blood Cell (RBC) Transfusions
Description: RBC transfusions could be given during the study, if medically necessary, i.e., in participants with severe anemia with distinct symptoms or signs of anemia (such as in participants with acute blood loss, with severe angina, or whose hemoglobin decreased to critical levels).
Time Frame: Baseline to Month 9
Population: ITT population
Measure: Number; unit: number of transfusions
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 178
number of transfusions | 39

ADVERSE EVENTS:
Time Frame: Baseline to Month 11
Description: Safety population
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Serious Adverse Events (participants affected / at risk) | 88/184
Other Adverse Events (participants affected / at risk) | 109/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-epoetin Beta (N=184)
Renal failure (Renal and urinary disorders) | 27
Renal failure chronic (Renal and urinary disorders) | 8
Renal impairment (Renal and urinary disorders) | 5
Renal failure acute (Renal and urinary disorders) | 2
Renal cyst haemorrhage (Renal and urinary disorders) | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 12
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 6
Anaemia (Blood and lymphatic system disorders) | 3
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1
Shunt occlusion (Injury, poisoning and procedural complications) | 5
Anaemia postoperative (Injury, poisoning and procedural complications) | 2
Drug toxicity (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1
Cardiac failure (Cardiac disorders) | 4
Angina unstable (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 2
Tachyarrhythmia (Cardiac disorders) | 2
Bradycardia (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Sepsis (Infections and infestations) | 3
Bronchitis (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes zoster ophthalmic (Infections and infestations) | 1
Meningitis enterococcal (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Drug ineffective (General disorders) | 2
Medical device complication (General disorders) | 2
Device dislocation (General disorders) | 1
Device malfunction (General disorders) | 1
Oedema (General disorders) | 1
Pyrexia (General disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Cachexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Diabetic foot (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Poor peripheral circulation (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
Haemoglobin decreased (Investigations) | 2
Blood pressure increased (Investigations) | 1
Blood sodium decreased (Investigations) | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Hypertensive encephalopathy (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1
Kidney transplant rejection (Immune system disorders) | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Retinal artery occlusion (Eye disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-epoetin Beta (N=184)
Vertigo (Ear and labyrinth disorders) | 13
Hyperparathyroidism secondary (Endocrine disorders) | 17
Nausea (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 12
Oedema (General disorders) | 28
Oedema peripheral (General disorders) | 20
Fatigue (General disorders) | 10
Bronchitis (Infections and infestations) | 11
Urinary tract infection (Infections and infestations) | 10
Iron deficiency (Metabolism and nutrition disorders) | 13
Hyperphosphataemia (Metabolism and nutrition disorders) | 11
Acidosis (Metabolism and nutrition disorders) | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13
Hypertension (Vascular disorders) | 56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.